CLINICAL TRIAL: NCT03452033
Title: A Phase 1/2a Randomized, Double-masked, Placebo Controlled, Dose-ranging Study of the Safety and Efficacy of H-1337 in Subjects With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension
Brief Title: H-1337 Ophthalmic Solution Phase 1/2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allysta Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALY337-201
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Glaucoma, Open-Angle
Keywords: glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Intervention Model Description: Double-masked, parallel
Who Masked: Participant, Investigator
Masking Description: Double-masked containers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- H-1337 Placebo (Placebo Comparator): H-1337 Placebo
  Interventions: Drug: H-1337 Placebo
- H-1337 [1] (Experimental): H-1337 [1]
  Interventions: Drug: H-1337 [1]
- H-1337 [2] (Experimental): H-1337 [2]
  Interventions: Drug: H-1337 [2]
- H-1337 [3] (Experimental): H-1337 [3]
  Interventions: Drug: H-1337 [3]

INTERVENTIONS:
Drug: H-1337 Placebo — H-1337 Placebo Vehicle
  Other Names: Vehicle
  Arms: H-1337 Placebo
Drug: H-1337 [1] — H-1337 Ophthalmic Solution Concentration 1
  Other Names: H-1337 conc 1
  Arms: H-1337 [1]
Drug: H-1337 [2] — H-1337 Ophthalmic Solution Concentration 2
  Other Names: H-1337 conc 2
  Arms: H-1337 [2]
Drug: H-1337 [3] — H-1337 Ophthalmic Solution Concentration 3
  Other Names: H-1337 conc 3
  Arms: H-1337 [3]

SUMMARY:
The study will evaluate the safety, tolerability, and preliminary efficacy of three concentrations of H-1337 and vehicle administered twice daily in a parallel group, double-masked design for 28 days of dosing in patients with elevated intraocular pressure (IOP).

DETAILED DESCRIPTION:
Study ALY337-201 will be a double-masked, randomized, placebo-controlled, dose-response study assessing the safety and ocular hypotensive efficacy of H-1337 ophthalmic solution in subjects with ocular hypertension (OHT) or open angle glaucoma.

During screening, subjects who meet the preliminary inclusion/exclusion criteria will discontinue use of their ocular hypotensive therapy during the washout period. The washout duration will be dependent on the subject's pre-study ocular hypotensive therapy. Starting on Day 0, those who continue to meet the inclusions/exclusion criteria and the diurnal IOP criteria will be randomized into one of the treatments arms and dosing will be initiated, continuing for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Diagnosis of bilateral primary open angle glaucoma or ocular hypertension.
3. One qualifying IOP criteria after washout:

   • Baseline (Day 0) at T0 (T0 = 8 am ± 30 min) IOP ≥ 23 mmHg in the study eye.
4. IOP criteria after washout ≤ 32 mmHg oculus uterque (OU) at all time points.
5. Best-corrected visual acuity (BCVA) in both eyes of 20/200 or better on Snellen, equivalent to + 1.0 log Mar.
6. Able and willing to sign informed consent, follow study instructions and complete all study visits.
7. As applicable, must be willing to discontinue the use of all ocular hypotensive medication(s) in both eyes prior to receiving the study medication and for the entire course of the study.
8. Able to self-administer or have a caretaker administer study eye drops.

Exclusion Criteria:

Ophthalmic:

Exclude subjects with:

1. Closed or very narrow angles (Grade 0-1) (see Section 5, gonioscopy) or those the investigator judges as occludable and/or with evidence of peripheral anterior synechiae (PAS) ≥ 180 degrees by gonioscopy within 6 months prior to Screening Visit in either eye. (Patent laser iridotomy with Grade 1-2 angles is acceptable in either eye, providing the PAS criteria are still met).
2. Previous glaucoma intraocular surgery in either eye. Prior laser trabeculoplasty (ALT or SLT) in either eye is allowed if performed more than 6 months prior to Screening Visit.
3. Any non-glaucoma intraocular surgery within 3 months prior to Screening Visit in either eye.
4. Intraocular laser surgery such as laser capsulotomy, laser iridotomy, and/or retinal laser within 1 month prior to Screening Visit in either eye.
5. Significant media opacity in either eye that would impede adequate posterior segment examination.
6. Contraindications to pupil dilation in either eye.
7. Other forms of glaucoma such as primary congenital, juvenile onset, chronic angle closure, and secondary glaucoma of any type including steroid-induced, inflammation-induced, or exfoliation glaucoma in either eye. Pigment dispersion syndrome/glaucoma is permitted in either eye.
8. Clinically significant corneal dystrophy, epithelial or endothelial disease, corneal irregularities or scarring that, in the investigator's judgment, would impede an accurate measurement of IOP or visualization of intraocular anatomy in the study eye.
9. History of refractive surgery in either eye (i.e., radial keratotomy, photorefractive keratectomy, LASIK).
10. History of corneal cross-linking procedure in either eye.
11. Unwillingness to be contact lens free during study participation.
12. Any history of uveitis, keratitis, or scleritis in either eye.
13. Any history of penetrating ocular trauma in either eye.
14. History within 3 months prior to Screening Visit of clinically significant moderate or severe chronic or active blepharitis, ocular dermatitis, or recent ocular conjunctivitis and/or ocular inflammation in either eye. Mild blepharitis, hyperemia (due to prostaglandin use) and/or blepharitis, and/or mild inactive seasonal allergic conjunctivitis and non-infective dermatitis are acceptable.
15. Corneal thickness < 480 or > 620 µm in the study eye. Pachymetry measurement within 6 months prior to Screening Visit is acceptable.
16. Advanced or severe glaucoma with progressive visual field loss and/or optic nerve changes in either eye that, in the investigator's best judgment, prevent safe withdrawal from treatment for the time periods required in this protocol.
17. Progressive retinal (including, but not limited to worsening dry age-related macular degeneration (AMD), presence of active wet AMD, or unstable diabetic retinopathy) or optic nerve disease in either eye from any cause other than glaucoma.
18. Any prior intravitreal steroid injection in either eye.
19. Sub-tenon's, sub-conjunctival or periocular steroid injections within the 6 months prior to Screening Visit in either eye.
20. Any use of ocular topical corticosteroids in either eye within 7 days, or chronic (as determined by the investigator) topical steroids within 28 days prior to Baseline and ensuing trial participation.
21. Known hypersensitivity to any component of the H-1337 formulation, including benzalkonium chloride, or to topical anesthetics or diagnostic drops used during the study.
22. Any ocular, condition that, in the investigator's judgment, could prevent the subject from safe participation the study.
23. Planned ocular surgery or intraocular injection procedure in either eye during study participation.

    General/Systemic:
24. Participation in a clinical study with use of any investigational drug or treatment within 30 days prior to Baseline (Day 0).
25. Clinically significant abnormalities in: laboratory tests, physical examination, vital signs and/or ECG at Screening Visit. If in the investigator's judgment a subject with clinically significant abnormalities is appropriate for enrollment in the study, a discussion between the investigator and the Medical Monitor must occur and be documented prior to enrollment of this subject in the study.
26. Clinically significant systemic, psychiatric or psychological disease (for example, renal, hepatic, uncontrolled diabetes, uncontrolled blood pressure, autoimmune disorders, psychiatric disorders, endocrine disorders, or any other disorders) or dependency which, in the investigator's judgment, would be unsafe and interfere with interpretation of the study results or the subject's ability to comply with the study requirements.
27. Anticipated changes or initiation of medications which might affect IOP and/or systemic blood pressure within 7 days prior to Baseline/Day 0 (e.g., oral anti-hypertensives such as sympathomimetic agents, beta-adrenergic blocking agents, alpha agonists, alpha adrenergic blocking agents, calcium channel blockers, angiotensin converting enzyme inhibitors; [diuretics are allowed]), and 2 months prior to Baseline/Day 0 for corticosteroids (i.e., oral, nasal, topical [dermal, mucosal], and/or inhaled corticosteroids). If there are no further anticipated changes in medications that could affect IOP and/or systemic blood pressure, then once the subject is stable on their new dose of medication for the required time period, the subject may complete the Baseline Visit, assuming that all other screening requirements are met. Medications used on an adjustable or sliding scale based on testing results are allowed.
28. Known history of Hepatitis B + C, HIV+, or AIDS and/or inadequate venous access.
29. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative serum pregnancy test result at Screening Visit and a negative urine and serum pregnancy test at Baseline (Day 0) prior to randomization in the study and must not intend to become pregnant during the study.
30. History of drug or alcohol abuse within the last 5 years.
31. Related to site study staff and/or site employees.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRN, Goose Creek, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan at current.

REFERENCES:
- [Derived] Hartman PJ, Cooke DL, Hsu HH, Stewart J, Sumi K, Yoshida Y, Hidaka H, Novack GD. Phase Ⅰ/Ⅱ, Double-Masked, Randomized, Vehicle-Controlled Study of H-1337 Ophthalmic Solution for Glaucoma and Ocular Hypertension. Ophthalmol Glaucoma. 2023 Mar-Apr;6(2):198-205. doi: 10.1016/j.ogla.2022.08.015. Epub 2022 Aug 31. PMID 36055467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 87 subjects were enrolled and randomized across 6 investigational sites in the United States.
Pre-assignment Details: During the screening phase (Screening and Baseline Visits), subjects washed out any current ocular hypotensive therapy according to the below schedule:
  Muscarinic agonists (eg, pilocarpine) and oral or topical carbonic anhydrase inhibitor (CAIs): ≥5 days Alpha adrenoceptor agonists: ≥5 weeks Beta-adrenoceptor antagonists: ≥6 weeks Prostaglandin analogues and combination drugs (use longest wash-out period of individual components): ≥6 weeks
Units Other Than Participants: study eyes
Groups:
- H-1337 0.06%: H-1337 Ophthalmic Solution Concentration 0.06%
- H-1337 0.2%: H-1337 Ophthalmic Solution Concentration 0.2%
- H-1337 0.6%: H-1337 Ophthalmic Solution Concentration 0.6%
- Vehicle: Vehicle (contains all components of the active formulation with the exception of H-1337)
Period: Overall Study
Arm/Group | H-1337 0.06% | H-1337 0.2% | H-1337 0.6% | Vehicle
Started | 21; 21 study eyes | 22; 22 study eyes | 22; 22 study eyes | 22; 22 study eyes
Completed | 21; 21 study eyes | 22; 22 study eyes | 22; 22 study eyes | 22; 22 study eyes
Not Completed | 0; 0 study eyes | 0; 0 study eyes | 0; 0 study eyes | 0; 0 study eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H-1337 0.06% | H-1337 0.2% | H-1337 0.6% | Vehicle | Total
Number analyzed (Participants) | 21 | 22 | 22 | 22 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (13.58) | 64.1 (10.02) | 67.4 (11.72) | 65.0 (14.44) | 64.5 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 14 | 12 | 52
  Male | 8 | 9 | 8 | 10 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 1 | 9
  Not Hispanic or Latino | 19 | 19 | 19 | 21 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 4 | 10
  White | 20 | 20 | 19 | 18 | 77
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 22 | 22 | 87
Intraocular pressure [Count of Participants; unit: Participants] — measured in mmHg
  Randomization stratum for IOP (≤26 mmHg and >26 mmHg)
  Participants
    ≤26 mmHg | 14 | 14 | 15 | 15 | 58
    >26 mmHg | 7 | 8 | 7 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Mean change in IOP from baseline on Day 28 (Time 0 + 4h)
Time Frame: Baseline and 28 days
Population: mmHg in the study eye
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: study eyes
Groups:
- H-1337 0.06%: H-1337 Ophthalmic Solution 0.06%
- H-1337 0.2%: H-1337 Ophthalmic Solution 0.2%
- H-1337 0.6%: H-1337 Ophthalmic Solution 0.6%
Arm/Group | H-1337 0.06% | H-1337 0.2% | H-1337 0.6% | Vehicle
Number analyzed (Participants) | 21 | 22 | 22 | 22
Number analyzed (study eyes) | 21 | 22 | 22 | 22
mm Hg | -4.45 (3.801) | -5.16 (3.114) | -4.93 (3.110) | -0.39 (2.355)

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | H-1337 0.06% | H-1337 0.2% | H-1337 0.6% | Vehicle
Number analyzed (Participants) | 21 | 22 | 22 | 22
Participants | 9 | 9 | 14 | 4

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | H-1337 0.06% | H-1337 0.2% | H-1337 0.6% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 9/21 | 9/22 | 14/22 | 4/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H-1337 0.06% (N=21) | H-1337 0.2% (N=22) | H-1337 0.6% (N=22) | Vehicle (N=22)
Eye disorders (Eye disorders) | 5 (21) | 3 (22) | 5 (22) | 2 (22)
General disorders and administration site conditiions (General disorders) | 6 (21) | 8 (22) | 13 (22) | 2 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03452033/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03452033/SAP_001.pdf